CLINICAL TRIAL: NCT03786159
Title: Prospective Nationwide Audit of the Management of Adhesive Small Bowel Obstruction: a Snapshot Study
Brief Title: National Snapshot Study Adhesive Small Bowel Obstruction (ASBO)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SnapshotASBO
Record Dates: First submitted 2018-11-30; First posted 2018-12-24 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2018-11

CONDITIONS: Surgery-Induced Tissue Adhesion; Surgical Adhesions; Adhesion, Tissue
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Over 63-90% of patients develop peritoneal adhesions after abdominal or pelvic surgery. Which makes it the most common complication after abdominal or pelvic surgery. Adhesions comprise a lifelong risk of adhesion related complications.The most frequent emergency complication of adhesion is an episode of adhesive small bowel obstruction (ASBO). Over 1 in 5 patients experiences at least 1 episode of ASBO in the 10 years following initial abdominal surgery. Despite the high incidence of ASBO, diagnosis and treatment of an episode of ASBO varies greatly between hospitals and even between doctors. Until now, optimal treatment patterns are unknown. The aim of this study is mapping of care for patients with a suspected episode of ASBO. With the collected data new hypothesis will be generated for the ideal diagnostic and therapeutic workflow for patients with a suspicion of an episode of ASBO.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion ASBO
* Age 18 years or older

Exclusion Criteria:

* Clear other cause of small bowel obstruction (e.g. tumor, hernia)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with a suspicion of ASBO, older than 17 years, can be included in the present snapshot study. Patients with an episode of small bowel obstruction that is certainly not caused by adhesions fall outside of the scope of this study (eg. tumor as cause of SBO).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
CT treatment ASBO | February 2021
  In how many patients does CT-scan impact initial management of ASBO (i.e. different cause of SBO found, or conservative trial vs. direct surgery)?
Diagnostics ASBO | February 2021
  How many patients in the Netherlands presenting with adhesive small bowel obstruction have a CT-scan in their diagnostic work-up?
Timeframe conservative trial ASBO | February 2021
  How long do Dutch surgeons continue a conservative trial in patients with persistent obstruction who are not clinically deteriorating? Outcome measures will be based on data from the online Case Report Form (CRF).
Conservative trial > 72 hours ASBO | February 2021
  Does continuing a conservative trial for more than 72 hours adverse impact final outcomes? Complications as measured by Clavien-Dindo will be registered and compared between groups.
Laparoscopic surgery for ASBO | February 2021
  How many patients that are surgically treated for ASBO in the Netherlands have laparoscopic surgery?
Outcome laparoscopic surgery for ASBO | February 2021
  What are the outcomes of laparoscopic surgery for ASBO? Days of in hospital stay, postoperative complications (Clavien-Dindo) and 90-day readmissions rates will be compared between patients who underwent open or laparoscopic surgery for ASBO.

CONTACTS AND LOCATIONS:
Overall Officials: Richard PG ten Broek, PhD, MD, Study Director — Radboudumc, departement of surgery
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ellis H, Moran BJ, Thompson JN, Parker MC, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Brien F, Buchan S, Crowe AM. Adhesion-related hospital readmissions after abdominal and pelvic surgery: a retrospective cohort study. Lancet. 1999 May 1;353(9163):1476-80. doi: 10.1016/S0140-6736(98)09337-4. PMID 10232313
- [Background] Parker MC, Ellis H, Moran BJ, Thompson JN, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Briena F, Buchan S, Crowe AM. Postoperative adhesions: ten-year follow-up of 12,584 patients undergoing lower abdominal surgery. Dis Colon Rectum. 2001 Jun;44(6):822-29; discussion 829-30. doi: 10.1007/BF02234701. PMID 11391142
- [Background] Luijendijk RW, de Lange DC, Wauters CC, Hop WC, Duron JJ, Pailler JL, Camprodon BR, Holmdahl L, van Geldorp HJ, Jeekel J. Foreign material in postoperative adhesions. Ann Surg. 1996 Mar;223(3):242-8. doi: 10.1097/00000658-199603000-00003. PMID 8604903
- [Background] Menzies D, Ellis H. Intestinal obstruction from adhesions--how big is the problem? Ann R Coll Surg Engl. 1990 Jan;72(1):60-3. PMID 2301905
- [Background] Diamond MP, Freeman ML. Clinical implications of postsurgical adhesions. Hum Reprod Update. 2001 Nov-Dec;7(6):567-76. doi: 10.1093/humupd/7.6.567. PMID 11727865
- [Background] Hershlag A, Diamond MP, DeCherney AH. Adhesiolysis. Clin Obstet Gynecol. 1991 Jun;34(2):395-402. doi: 10.1097/00003081-199106000-00023. PMID 1831077
- [Background] Beck DE, Opelka FG, Bailey HR, Rauh SM, Pashos CL. Incidence of small-bowel obstruction and adhesiolysis after open colorectal and general surgery. Dis Colon Rectum. 1999 Feb;42(2):241-8. doi: 10.1007/BF02237135. Erratum In: Dis Colon Rectum 1999 May;42(5):578. PMID 10211502

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03786159/Prot_SAP_000.pdf